CLINICAL TRIAL: NCT05915026
Title: A Multicenter, Prospective, Open-label Study to Evaluate the Pharmacokinetics and Safety of Gadoquatrane in Pediatric Participants (From Birth to <18 Years) Undergoing Contrast-enhanced Magnetic Resonance Imaging (CE-MRI)
Brief Title: A Study to Learn How Gadoquatrane Moves Into, Through, and Out of the Body and How Safe it is in Children (From Birth to <18 Years), Who Will Undergo a Contrast Enhanced MRI (Quanti Pediatric)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21196; 2022-501883-17-00 (Other: CTIS (EU))
Record Dates: First submitted 2023-06-14; First posted 2023-06-22 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gadoquatrane (Experimental): Participants will receive one intravenous injection of gadoquatrane during MRI.
  Interventions: Drug: Gadoquatrane (BAY1747846)

INTERVENTIONS:
Drug: Gadoquatrane (BAY1747846) — 0.04 mmol Gd/kg body weight, solution for intravenous injection, single dose

SUMMARY:
Researchers are looking for a better way to help children under the age of 18 with any known or suspected problems scheduled for a "contrast-enhanced" Magnetic Resonance Imaging (MRI).

MRI is used by doctors to create detailed images of the inside of the body to identify health problems. Sometimes doctors need to inject a contrast agent into a patient's vein to perform a "contrast-enhanced" MRI (CE-MRI). Such CE-MRI examinations may support doctors to identify certain health problems or improve their evaluation.

The contrast agents commonly used in MRI are gadolinium-based contrast agents (GBCAs). GBCAs contain a "rare earth" element called gadolinium (Gd), which is needed for the increase in signal intensity and contrast in MRI. The gadolinium in these contrast agents is caged in a molecule (chelate complex). Researchers are developing new contrast agents with a lower amount of Gd needed per CE-MRI investigation. Gadoquatrane is one of these new contrast agents. It has been tested in several studies previously.

The main purpose of this study is to learn how gadoquatrane moves into, through, and out of the body and how safe it is in children. The researchers will measure the amount of gadoquatrane in the blood at different time points after a single injection.

The participants will undergo an MRI examination and receive gadoquatrane once at a dose of 0.04 mmol Gd/kg (corresponding to 0.1 mL/kg). It is injected into the participant's vein (also called an intravenous injection) during the MRI examination.

Each participant will be in the study for between 8 and 38 days with up to 5 doctor visits, including the screening phase of up to 28 days with no more than 2 visits. Once a participant has received the injection of gadoquatrane, the remaining study duration is 7 (±1) days.

At the start or during the study, the doctors and their study team will:

* check the weight and height of the participant,
* ask for information including age and medical history,
* take participants' blood samples,
* ask participants and/or their guardians questions about medicines they are taking,
* check blood pressure, heart rate and body temperature,
* check the area where the participants had the intravenous injection,
* do pregnancy tests in girls of childbearing age,
* review the MRI scans obtained in the study and decide on the diagnosis
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants from birth to <18 years of age at the time of signing the informed consent form.
* Participants who have a clinical indication to undergo a CE-MRI for any clinical condition in any body region and who can undergo study procedures as per Investigator judgement.
* Participants can be male or female (according to their reproductive organs and functions assigned by chromosomal complement).
* Female contraception and barriers as well as pregnancy testing is required as appropriate for the age and sexual activity of pediatric participants and as required by local regulations.
* The legal guardian(s) is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* When applicable by law for a participant, a legal guardian must be available to help the study-site personnel ensure follow up, accompany the participant to the study site on each assessment day, and consistently and consecutively be available to provide information on the participant during the scheduled study visits.

Exclusion Criteria:

* Body weight <2500 g at screening and baseline
* The medical condition and/or local allowance for maximum blood draw in the pediatric participant is not suitable for study procedures, including pharmacokinetics (PK) and safety blood draws, without compromising any expected clinical care/procedure need.
* Acute kidney injury (i.e., acute renal failure).
* Age-adjusted renal function is "decreased" (eGFR <80% of age adjusted normal renal function) as evaluated by the investigator based on a serum or plasma creatinine result obtained within 2 weeks prior to study intervention.
* Considered clinically unstable or has a concurrent/concomitant condition that may not allow participation for the full planned study period, in the judgement of the investigator.
* History of moderate to severe allergic-like reaction to any GBCA.
* Bronchial asthma considered unstable or had major therapeutical modification within last 4 weeks.
* Severe cardiovascular disease, except for cardiac or vascular magnetic resonance (MR), if considered clinically justified by the investigator.
* Planned or expected intervention (e.g., treatment or procedure) or change in treatment (e.g. start of chemotherapy) that may significantly affect study parameters (i.e. safety/adverse events [AEs] [e.g. confounding AEs or safety events due to surgery or chemotherapy], PK parameters) or would prevent the participant from performing study procedures, from the administration of gadoquatrane up to the 24 h ± 4 h follow-up.
* Participants who received or will receive any other contrast agent within 72 hours prior to gadoquatrane injection or up to 72 hours after gadoquatrane injection.
* Contraindications to the administration of GBCAs (depending on local product label), or history of adverse reaction to GBCAs.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of gadoquatrane after single administration | Up to 8 hours post injection
Plasma clearance normalized to body weight (CL/BW) of gadoquatrane after single administration | Up to 8 hours post injection
Apparent volume of distribution at steady state normalized to body weight (Vss/BW) of BAY1747846 after single administration | Up to 8 hours post injection
Simulation of plasma concentration at 20 min post-injection (C20) | At 20 minutes post injection

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events, including serious adverse events | Within 24 (± 4) hours post injection
Number of participants with treatment emergent adverse events, including serious adverse events, per intensity | Within 24 (± 4) hours post injection
Number of participants with post-treatment adverse events, including serious adverse events | Up to 7 (± 1) days after the day of study intervention
Number of participants with post-treatment adverse events, including serious adverse events, per intensity | Up to 7 (± 1) days after the day of study intervention

CONTACTS AND LOCATIONS:
Locations (34):
- United States (3):
  - Halo Diagnostics - Indian Wells, Indian Wells, California
  - Children's Mercy Hospital Kansas City - Radiology, Kansas City, Missouri
  - MUSC University Hospital - Radiology, Charleston, South Carolina
- Argentina (3):
  - Centro de Diagnostico Enrique Rossi | Departamento de Investigacion Clínica, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Sanatorio Allende | Departamento de Investigación Clínica, Córdoba
  - Clinica Universitaria Reina Fabiola | Consultorios Externos, Córdoba
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment Sveti Georgi | Base II - Radiology Department, Plovdiv
  - Multiprofile Hospital for Active Treatment Central Onco Hospital | Independent Medical Diagnostic Laboratory Mediscan, Plovdiv
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski | Radiology Department, Sofia
  - University Hospital for Active Treatment Tsaritsa Joanna - ISUL | Radiology Department, Sofia
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada
- China (4):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Children's Hospital Zhejiang University School of Med, Hangzhou, Hangzhou Province
  - West China Second University Hospital, Chengdu, Sichuan
- Czechia (2):
  - Fakultní nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
- Germany (5):
  - Universitätsklinikum Münster - Klinik für Radiologie, Kinderradiologie, Münster, North Rhine-Westphalia
  - Universitätsklinikum Leipzig - Institut für Kinderradiologie, Leipzig, Saxony
  - Universitätsklinkum Halle (Saale) - Universitätsklinik und Poliklinik für Radiologie, Kinderradiologie, Halle, Saxony-Anhalt
  - Universitätsklinikum Jena - Institut für Diagnostische und Interventionelle Radiologie, Kinderradiologie, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Pädiatrische Radiologie, Berlin
- Japan (10):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo, Tokyo
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Nara Prefecture General Medical Center, Nara
  - Shizuoka Children's Hospital, Shizuoka
- Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw, Poland
- Karolinska Universitetssjukhuset Solna - Funktion Medicinsk Diagnostik, Barnradiologi, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.